CLINICAL TRIAL: NCT03453827
Title: Assessment of Long-term Intraocular Lens (IOL) Decentration and Tilt in Eyes With Pseudoexfoliation Syndrome (PES) Following Cataract Surgery
Brief Title: Long-term Intraocular Lens (IOL) Decentration and Tilt in Eyes With Pseudoexfoliation Syndrome (PES) Following Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Hospital Hietzing (Other)
Responsible Party: Principal Investigator, Kata Mihaltz, Oberarzt M.D. PhD FEBO, Hospital Hietzing
Other Study IDs: PEX Study
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Cataract; Pseudoexfoliation Syndrome; Pseudophakia
Keywords: Pseudoexfoliation Syndrome; Cataract; Aberration; IOL decentration; IOL tilt
MeSH Terms: conditions — Cataract; Exfoliation Syndrome; Pseudophakia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEX: Patients after Cataract surgery with PES
  Interventions: Other: no intervention
- Control: Patients after Cataract surgery without PES
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
To evaluate long-term intraocular lens (IOL) decentration and tilt in eyes with pseudoexfoliation syndrome (PES) following cataract surgery using Visante anterior segment OCT and iTrace Visual Function Analyzer.

DETAILED DESCRIPTION:
64 eyes following cataract surgery from 2009 to 2012 were included, 34 eyes had PES, 30 eyes did not show PES. A standard phacoemulsification procedure followed by IOL implantation was performed and patients were followed 4-6 years after surgery (mean=69 months). Best corrected visual acuity (BCVA), intraocular pressure (IOP) and capsulorhexis size were measured. IOL tilt and IOL decentration were evaluated using Visante Omni anterior segment OCT (Carl Zeiss Jena GmBH, Germany). The iTrace VFA (Visual Function Analyzer, Topcon Medical Systems, Inc.) was used to measure internal, corneal and total optical aberrations.

ELIGIBILITY:
Inclusion Criteria:

* patients 4-6 years after standard cataract surgery
* pseudoexfoliation Syndrome (PES)

Exclusion Criteria:

* Diabetic retinopathy
* Age related macula Degeneration
* retinal bloodvessel disease

Ages: 18 Years to 125 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent standard procedure cataract surgery with or without Pseudoexfoliation Syndrome.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
IOL decentration | 4-6 years after cataract surgery
  decentration of IOL is measured using Hoya iTrace
IOL tilt | 4-6 years after cataract surgery
  tilt of implanted IOL is measured using Hoya iTace
IOL decentration | 4-6 years after cataract surgery
  decentration of IOL is measured using Zeiss OCT
IOL tilt | 4-6 years after cataract surgery
  tilt of implanted IOL is measured using Zeiss OCT